CLINICAL TRIAL: NCT01776151
Title: Arterial Elasticity: A Substudy of Strategic Timing of AntiRetroviral Treatment (START)
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0603M83587-3
Record Dates: First submitted 2012-09-18; First posted 2013-01-25 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; HIV
Keywords: HIV; cardiovascular diseases; vascular stiffness
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Citrated plasma is collected at each study visit and stored at a central lab for future assessment of changes in plasma markers of thrombosis and fibrinolysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out if starting anti-retroviral therapy (ART) above 500 cluster-of-differentiation-4 (CD4)+ cells/milliliter (mL) ('early ART group') is better at reducing the stiffness of arteries than waiting to start ART until the CD4+ drops below 350 cells/mL ('deferred ART group'). Artery stiffness has been associated with an increased risk of cardiovascular (heart) disease, and could be useful as an earlier indicator of heart disease. In this study, the stiffness of arteries will be measured at study entry, months 4, 8, 12, and annually thereafter, using a tonometer on the participant's forearm.

ELIGIBILITY:
Inclusion Criteria:

* Simultaneous co-enrollment in the START study
* Signed informed consent

Exclusion Criteria:

* Inability to ascertain waveform measurements that can be analyzed, i.e. atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollees are HIV-positive, antiretroviral-naive individuals with CD4+ > 500 cells/mL randomized to the START trial.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in large artery elasticity (LAE | baseline, Months 1, 4, 8, 12, annually thereafter
  Large artery elasticity is measured using a tonometer placed on the forearm.
Change from baseline in small artery elasticity (SAE) | baseline, Months 1, 4, 8, 12, annually thereafter
  Small artery elasticity is measured using a tonometer placed on the forearm.

SECONDARY OUTCOMES:
Changes in plasma markers of thrombosis and fibrinolysis | baseline, months 4, 8, 12, annually thereafter
  Citrated plasma will be collected and stored for central measurement of plasma markers of thrombosis and fibrinolysis in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Jason V Baker, MD, Study Chair — University of Minnesota; Daniel Duprez, MD, PhD, Study Chair — University of Minnesota
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Derived] Baker JV, Engen NW, Huppler Hullsiek K, Stephan C, Jain MK, Munderi P, Pett S, Duprez D; International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) START Study Group. Assessment of arterial elasticity among HIV-positive participants with high CD4 cell counts: a substudy of the INSIGHT Strategic Timing of AntiRetroviral Treatment (START) trial. HIV Med. 2015 Apr;16 Suppl 1(0 1):109-18. doi: 10.1111/hiv.12239. PMID 25711329
- See also: INSIGHT network website, including information on the START Arterial Elasticity Substudy — http://www.insight-trials.org